CLINICAL TRIAL: NCT06756386
Title: Effect of Extra Corporeal Shock Wave Versus Low Level Laser on Chronic Venous Ulcer Healing
Brief Title: Shock Wave Versus Low Level Laser on Chronic Venous Ulcer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mahmoud Awad Ramadan Elkholy, Lecturer of Physical Therapy for Integumentary System and burn disorders, Faculty of Physical Therapy ,Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/02012024/AHMED
Record Dates: First submitted 2024-12-13; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Venous Ulcer
Keywords: shock wave , low level laser
MeSH Terms: conditions — Varicose Ulcer | interventions — Low-Level Light Therapy; Conservative Treatment

STUDY DESIGN:
Intervention Model Description: 1. study group (A) include old age patients with venous ulcer will receive extra corporeal shock wave therapy along with conservative treatment (compression therapy (pressure garment),lifestyle changes, physical activity) plus medical treatment
  2. study group (B) include old age patient with chronic venous ulcer will receive low level laser therapy along with conservative treatment (compression therapy (pressure garment), lifestyle changes,physical activity) Plus medical treatment
  3. control group (C) include old age patients with venous ulcers will receive conservative treatments ( compression pandaging, lifestyle changes, physical activities) plus medical treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group A (Active Comparator): study group (A) include 15 old age patients with venous ulcer will receive extra corporeal shock wave therapy along with conservative treatment (compression therapy (pressure garment),lifestyle changes, physical activity) plus medical treatment
  Interventions: Device: extra corporeal shock wave therapy (ESWT )
- Group B (Active Comparator): study group (B) include 15 old age patient with chronic venous ulcer will receive low level laser therapy along with conservative treatment (compression therapy (pressure garment), lifestyle changes,physical activity) Plus medical treatment
  Interventions: Device: Low Level Laser Therapy
- Group C (Active Comparator): control group (C) include 15 old age patients with venous ulcers will receive conservative treatments ( compression pandaging, lifestyle changes, physical activities) plus medical treatment
  Interventions: Other: conservative treatments

INTERVENTIONS:
Device: extra corporeal shock wave therapy (ESWT ) — Using wound area measurements and histological/immunohistochemical analysis of wound biopsies, we show ESWT enhanced healing of chronic ulcers associated with improved wound angiogenesis ), significantly decreased-positive macrophages per biopsy area and generally increased macrophage activity ,this activity prevent bacterial infection which delay healing
  Arms: group A
Device: Low Level Laser Therapy — Low-level laser therapy (LLLT) has been used as an adjuvant to conventional therapy with promising results,improve healing by delivering nutrient substances , especially in patients with acute and bloody ulcers.
  Positive effects include acceleration of tissue repair, increased formation of granulation tissue, wound contraction, inflammation modulation, and pain reduction The biochemical effects of LLLT are associated with the release of preformed substances (histamine, serotonin, and bradykinin), which stimulate the production of ATP and inhibit the production of prostaglandins.
  Arms: Group B
Other: conservative treatments — ( compression pandaging, lifestyle changes, physical activities)
  Arms: Group C

SUMMARY:
To find out the difference in the effect of shock wave therapy and low level laser therapy on venous ulcer patient As regards the following outcomes;

1. medical state of patient no ( diabetes, hypertension,obesity,cancer , rheumatoid)
2. The degree of ulcer
3. recurrence of ulcer
4. The degree of pain and disabilities
5. inflammatory marker

DETAILED DESCRIPTION:
45 venous ulcer patient of both sexes will be recruited in this study from cardiovascular units in nasser institute hospital , their age ranged from 45 to 60 years old and randomly divided into 3 equal groups

1. study group (A) include old age patients with venous ulcer will receive extra corporeal shock wave therapy along with conservative treatment (compression therapy (pressure garment),lifestyle changes, physical activity) plus medical treatment
2. study group (B) include old age patient with chronic venous ulcer will receive low level laser therapy along with conservative treatment (compression therapy (pressure garment), lifestyle changes,physical activity) Plus medical treatment
3. control group (C) include old age patients with venous ulcers will receive conservative treatments ( compression pandaging, lifestyle changes, physical activities) plus medical treatment The study will be conducted when the patient stable medically and will be conducted until complete healing of ulcer

ELIGIBILITY:
Inclusion Criteria:

* All old age patients will be
* Ranging from 45-60 years old
* With BMI from (25-30)
* Chronic venous ulcer grade 2 or 3
* Ulcers non infected with superficial blood insufficiency
* open ulcers.

Exclusion Criteria:

* -Diabetes
* hypertension
* rheumatoid arthritis
* Obesity
* Musculoskeletal disorders
* Dementia
* cerbrovascular stroke
* Deep venous thrombosis
* deep venous ulcer
* venous ulcer grade 4
* smokers

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
ulcer size | 4 weeks
  Smart phone application imito wound application was found to be reliable for three-dimensional analysis such as depths and volumes, its results were less suited for immediate application to clinical environments. .

SECONDARY OUTCOMES:
Venous Insufficiency Epidemiological and Economic Study - Quality of Life/Symptoms questionnaire | 4 weeks
  Veines questionnaire is a disease-specific quality of life instrument for chronic venous disorders of the leg .the responeses are rated on 2-point to 7- point response scales of intensity ,frequency, or agreement.These summary scores are transformed to T scores (mean, 50; standard deviation, 10) for easy interpretation.
  Participants whose ulcers had healed showed greater mean increase in scores than did those yet to heal, though they continued to report leg problems. An intrinsic scoring method appeared superior to the original relative method.
  VEINES-QOL was suitable for use in the study of venous leg ulcers. The intrinsic scoring method should be adopted, to facilitate comparisons between studies

IPD SHARING:
Plan to Share IPD: Undecided
university ethics

REFERENCES:
- [Background] Bavaresco T, Pires AUB, Moraes VM, Osmarin VM, Silveira DT, Lucena AF. Low-level laser therapy for treatment of venous ulcers evaluated with the Nursing Outcome Classification: study protocol for a randomized controlled trial. Trials. 2018 Jul 12;19(1):372. doi: 10.1186/s13063-018-2729-x. PMID 30001202
- [Background] Cooper B, Bachoo P. Extracorporeal shock wave therapy for the healing and management of venous leg ulcers. Cochrane Database Syst Rev. 2018 Jun 11;6(6):CD011842. doi: 10.1002/14651858.CD011842.pub2. PMID 29889978